CLINICAL TRIAL: NCT05084170
Title: Cingulotomy for Refractory Neuropathic Pain Following Spinal Cord Injury
Brief Title: Cingulotomy for Refractory Neuropathic Pain Following Spinal Cord Injury (CRNP-SCI)
Acronym: CRNP-SCI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: St George's, University of London (Other)
Responsible Party: Sponsor
Other Study IDs: 2021.0050
Record Dates: First submitted 2021-09-17; First posted 2021-10-19 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-10

CONDITIONS: Spinal Cord Injuries; Neuropathic Pain
MeSH Terms: conditions — Spinal Cord Injuries; Neuralgia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Bilateral anterior cingulotomy — Stereotactic bilateral anterior cingulotomy is a brain operation with demonstrated efficacy in the treatment of intractable pain from a variety of causes, including a few cases of spinal cord injury related neuropathic pain.

SUMMARY:
Neuropathic pain is very common following a spinal cord injury, estimated to affect 43% of patients after 6 months. A proportion of these patients do not respond to treatment and there remains an unmet need to treat people with refractory spinal injury related neuropathic pain. While neuropathic pain medications, baclofen pumps and spinal cord stimulation work for some patients, a significant number are refractory to these therapies. Chronic pain can contribute to loss of functional ability, mental health problems, and a worse quality of life.

Studies of functional neuroimaging have shown that the Anterior Cingulate Cortex (ACC) is a key structure in human pain perception, being part of a central pain neuromatrix or medial pain system, which includes thalamic nuclei and periaqueductal grey matter. A similar neuromatrix also including the insula is involved in the regulation of the autonomic nervous system, which explains the well-recognized interactions between pain and autonomic function. Moreover, it has been shown that the ACC is important for the emotional experience and thus the subjective intensity of pain, and it has a role in cognitive control processes for optimizing behaviour in the presence of pain.

Bilateral anterior cingulotomy has been demonstrated to be a safe and effective therapeutic option for patients with otherwise intractable pain syndromes of different origins, e.g., refractory pain due to cancer or stroke.

Although, cingulotomy has been shown to be a viable option in intractable pain of different origins, there remains a lack of evidence in patients with spinal cord injury and only scanty data are available in literature. Moreover, the effects of cingulotomy on mood, emotion processing, cognition and autonomic reactivity are not clear.

DETAILED DESCRIPTION:
Neuropathic pain is very common following spinal cord injury, with significant long-term impact on an individual's quality of life, functional ability and mental health, as well as increased utilisation of health care resources.

People living with the effects of spinal cord injury frequently suffer chronic neuropathic pain. A proportion of these do not respond to treatment and there remains an unmet need to treat people with refractory spinal injury related neuropathic pain. While spasms can be treated by baclofen pumps and neuropathic pain sometimes treated by spinal cord stimulation, many patients remain refractory to those surgical treatments. The research aims to establish the efficacy of bilateral anterior cingulotomy to treat chronic pain in people with spinal cord injury.

Stereotactic bilateral anterior cingulotomy is a brain operation with demonstrated efficacy in the treatment of intractable pain from a variety of causes, including a few cases of spinal cord injury related neuropathic pain. This may therefore be a therapeutic option for patients refractory to other treatments.

Significant recent advances in surgical and imaging techniques have vastly improved the outcomes and safety profile of stereotactic lesioning for multiple indications, most commonly movement disorders but also other conditions including pain.

However, only scanty epidemiological data on the effect of this procedure in people with chronic pain are available in the scientific literature so far and it is unclear the number of patients who may benefit from such a treatment. Few case reports have been published reporting a good outcome of bilateral cingulotomy on pain in patients with SCI [8]. Therefore, there is a hope that this procedure may offer significant relief and thus improved quality of life for a proportion of patients with SCI who have exhausted other treatment options.

The results of this open label study will provide important information on whether bilateral anterior cingulotomy is an effective treatment in improving pain refractory to other routinely offered treatments in patients with spinal cord injury. This will give scientific evidence for offering this procedure to these patients and alleviate their symptoms and improve their quality of life. If efficacy is established, it may become an established viable option in routine clinical practice.

The investigators aim to recruit 12 patients over a period of 24 months with 12 months' follow-up and to analyse and publish their results in the following 12 months. The investigators will ensure that findings will promptly reach the widest audience of potential beneficiaries (academic, clinical, patients and public audiences) to have a practical impact on clinical management of patients with SCI.

The investigators aim to demonstrate whether this procedure can provide sustained symptomatic relief while carefully monitoring for the development of adverse effects. They propose a pilot open label study of 12 patients with refractory neuropathic pain associated with spinal cord injury to determine the safety and efficacy of this procedure in this group of patients. The anterior cingulate cortex is involved not only in the regulation of pain but also in emotional and autonomic nervous system regulation, which the investigators will monitor closely to determine the nature of any effects that this procedure might cause.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of complete or partial spinal cord injury at any level
* Chronic neuropathic pain (for at least 12 months) resistant to conventional treatments or history of unacceptable side effects from conventional treatments.
* Age limits 18-70 years old

Exclusion Criteria:

* Traumatic brain injury
* Severe cognitive impairment
* Significant medical co-morbidity (e.g. coagulopathy)
* Radiofrequency lesioning or MRI incompatible device (e.g. baclofen pump or spinal cord stimulator) already in situ

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with neuropathic pain secondary to spinal cord injury, refractory to analgesia and other pain interventions
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2023-04-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
The primary outcome will be a change in pain scores (Neuropathic pain scale and Spinal cord injury pain inventory scores) at 3 and 12 months. | 12 months

SECONDARY OUTCOMES:
Improvement in health-related quality of life as measured by EuroQol 5 Dimension questionnaire. | 12 months
Connectomic changes in brain pain networks as assessed by magnetic resonance imaging. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Erlick Pereira, Study Chair — St George's, University of London
Locations (1):
- St. George's, University of London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No